CLINICAL TRIAL: NCT06765239
Title: Evaluation of Breathe-Easy Hayfever Care for Managing Symptoms in Patients With Seasonal Allergic Rhinitis
Brief Title: Breathe-Easy: Hayfever Care for Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innowage Limited (Industry)
Collaborators: Mettle Networks (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: InnUK/MN/0120
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hayfever; Allergy Pollen; Allergic Rhinitis
Keywords: Breathe-Easy; Hayfever Care
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hayfever Care (Experimental): Hayfever Care, a powdered natural food supplement.
  Interventions: Dietary Supplement: Hayfever Care
- Wait-list Care (Other): No supplement was given during the trial period
  Interventions: Other: Wait-list Control

INTERVENTIONS:
Dietary Supplement: Hayfever Care — Powdered natural food supplement provided as a decoction, to be taken twice daily.
  Personalized Diet and Nutrition Guidance along with Lifestyle Advice
  Other Names: Mettle's Hayfever Care
  Arms: Hayfever Care
Other: Wait-list Control — Personalized Diet and Lifestyle Advice
  Arms: Wait-list Care

SUMMARY:
This waitlist-controlled trial aims to evaluate the therapeutic effectiveness of Hayfever Care by assessing disease-specific symptoms over a 4-week period. Additionally, the study examines the tolerability and safety of the solution.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate symptoms during the hayfever season
* Generally healthy individuals without chronic illnesses
* Willingness to comply with study requirements, including completing symptom diaries.

Exclusion Criteria:

* History of anaphylaxis or severe hayfever symptoms requiring emergency treatment.
* Pregnant or breastfeeding
* History of substance abuse or excessive alcohol consumption.
* Use of systemic corticosteroids, immunotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Well-being Numerical Rating Scales | Change from Baseline to 4 weeks after baseline

SECONDARY OUTCOMES:
Change of Symptom Dry Eyes | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Itching Eyes | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Burning Eyes | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Respiratory Complaints | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Sneezing | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Rhinitis | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Fatigue | Change in symptom scores from baseline to 4 weeks.
Change of Symptom Headache | Change in symptom scores from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Shinde, Study Chair — Mettle Networks; Dr. Pradyuman S Rathore, Study Director — Innowage, India; Dr Mridu Sharma, Principal Investigator — Gyansanjeevani India
Locations (1):
- Gyansanjeevani India, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided